CLINICAL TRIAL: NCT06594094
Title: An Investigator-initiated Clinical Study Evaluating the CRISPR-hfCas12Max Gene Editing Therapy in the Treatment of Duchenne Muscular Dystrophy (DMD)
Brief Title: An Open-label, Multidose Dose-escalation Study to Understand the Safety of CRISPR Gene-editing Therapy and Its Long-Lasting Effects in DMD Patients (MUSCLE)
Acronym: MUSCLE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: HuidaGene Therapeutics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HG30201
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Duchenne Muscular Dystrophin (DMD)
Keywords: DMD; dystrophin; Gene-editing; HG302; CRISPR
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Intervention Model Description: Two dosing cohort:
  Low dose :2~3 subjects High dose: 2~3 subjects
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- HG302 (Experimental): The study will enroll up to 2 dose cohorts
  Interventions: Genetic: HG302

INTERVENTIONS:
Genetic: HG302 — Once intravenous injection; The duration of the study is about 32 weeks for each subject, including a 6 weeks screening period, enrollment visit, treatment visit, and 26 weeks follow-up period.

SUMMARY:
Duchenne muscular dystrophin (DMD) is an X-linked, fatal muscle-wasting disease caused by mutations in the DMD gene encoding the dystrophin proteins, with symptom onset before age of 6 years in boys. These mutations abolish dystrophin production in the muscle, leading to dystrophin deficiency at the myofiber membrane, continued fiber degeneration, the need for assisted ventilation, respiratory inflammation, loss of walking ability in their teens, followed by respiratory and cardiac decline, and eventually premature death before the age of 30.

Currently, there are only glucocorticoids for the standard supportive therapy of DMD, which can improve disease symptoms but do not change the outcome of the disease, Three antisense oligonucleotide (ASOs) medicines have been approved to treat DMD with exon 45-55 hotspot region mutations. However, they can only restore trace amounts of dystrophin protein, which is insufficient to bring real clinical benefits. Gene replacement therapy has been approved using adeno-associated virus (AAV) vectors to deliver the "mini-dystrophin" gene. Yet, mini-dystrophin gene-expression versions of truncated dystrophin functionality are sacrificed and limited.

HG302 uses a single AAV vector to deliver the CRISPR/hfCas12Max DNA editing system in the human DMD exon 51 splice donor site. Preclinical studies have shown that a single intravenous injection of HG302 significantly restores dystrophin protein expression in muscle fibers and rescues their muscle function in humanized DMD mice to wild-type levels, with long-lasting and durable efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Males ≥ 4 and ≤8 years at the time of signing informed consent, with clinical diagnosis of DMD;
* DMD gene mutation types are deletions in exons 52, 52-61, or 52-63;
* Able to walk at least 10 meters independently;
* Willing to cooperate with muscle biopsy test;
* Acceptable hematology, clinical chemistry, and urine laboratory parameters.

Exclusion Criteria:

* Presence of active infection;
* Presence of DMD-associated cardiomyopathy manifestations;
* Respiratory insufficiency requiring invasive or non-invasive ventilation;
* Serious infections such as pneumonia, pyelonephritis, or meningitis within 4 weeks prior to receiving trial drug infusion;
* Prior central nervous system surgery within 6 months before enrolment;
* Use of any investigational drug, or exon-skipping drug (whether investigational or not) 6 months prior to Screening;
* Previous treatment with any gene therapy or cell therapy (e.g., stem cell transplantation);
* Any other conditions that would not allow the potential subject to complete follow-up examinations during the study and would, in the opinion of the investigator, make the potential subject unsuitable for the study.

Ages: 4 Years to 8 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Estimated)
Dates: Start 2024-11-06 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of systemic adverse events | 26 weeks
  Number of adverse events (AEs), serious adverse events (SAEs), and dose-limiting toxicities (DLTs)

SECONDARY OUTCOMES:
Change from baseline in percentage of dystrophin positive fiber | 26 weeks
  Test percentage of dystrophin positive fiber to detection of dystrophin expression
Change from baseline in dystrophin fiber intensity | 26 weeks
  Test dystrophin fiber intensity to detection of dystrophin expression
Change from baseline in North Star Ambulatory Assessment scale | 26 weeks
  North Star Ambulatory Assessment scale documents motor performance in children, with total score range from 0-34, the higher score means better motor performance

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — HuidaGene Therapeutics Co., Ltd.
Locations (1):
- Shanghai Children s Medical Center Affiliated to Shanghai Jiao Tong University School of Medical, Shanghai, Shanghai Municipality, China